CLINICAL TRIAL: NCT06001151
Title: Cadonilimab (AK104) Plus Chemotherapy as First-line Treatment in Non-squamous Non-Small Cell Lung Cancer (NSCLC) Patients With Programmed Cell Death Ligand 1 (PD-L1) Negative：A Multi-center, Single-arm, Phase II Study
Brief Title: Cadonilimab (AK104) Plus Chemotherapy as First-line Treatment in Non-squamous Non-Small Cell Lung Cancer (NSCLC) Patients With Programmed Cell Death Ligand 1 (PD-L1) Negative
Acronym: ACHELOUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qian Chu (Other)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor-Investigator, Qian Chu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S019
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: non-squamous Non-Small Cell Lung Cancer; Programmed Cell Death Ligand 1; cadonilimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Patients will receive cadonilimab (10mg/kg) plus pemetrexed(500mg/m2) and carboplatin (AUC=5) every 3 weeks for 4 cycles, follwed with cadonilimab (10mg/kg) plus pemetrexed (500mg/m2) every 3 weeks as maintenance therapy.
  Interventions: Drug: Cadonilimab; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Cadonilimab — Patients receive cadonilimab (10mg/kg) every 3 weeks.
  Other Names: AK104
Drug: Pemetrexed — Patients receive pemetrexed (500mg/m2) every 3 weeks.
Drug: Carboplatin — Patients receive carboplatin (AUC=5) every 3 weeks for 4 cycles.

SUMMARY:
This is a single arm, multi-center clinical trial. Target population is advanced or metastatic non-squamous Non-Small Cell Lung Cancer (NSCLC) Patients with Programmed Cell Death Ligand 1 (PD-L1) negative, aiming to evaluate the efficacy and safety of the combination therapy of Cadonilimab and chemotherapy. Cadonilimab is a PD-1/CTLA-4 bi-specific antibody.

DETAILED DESCRIPTION:
This trial enrolled advanced or metastatic non-squamous Non-Small Cell Lung Cancer (NSCLC) Patients with Programmed Cell Death Ligand 1 (PD-L1) negative. Patients will receive cadonilimab (10mg/kg) plus pemetrexed(500mg/m2) and carboplatin (AUC=5) every 3 weeks for 4 cycles, follwed with cadonilimab (10mg/kg) plus pemetrexed (500mg/m2) every 3 weeks as maintenance therapy. The primary endpoint is 12-month progression-free-survival (PFS) rate assessed by investigators. Key secondary endpoints include objective response rate (ORR), duration of response (DOR), disease control rate (DCR), time to response (TTR), progression free survival (PFS), overall survival (OS), and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically/cytologically stage IIIB, IIIC, IV non-squamous Non-Small Cell Lung Cancer (NSCLC)
* PD-L1 TPS<1%
* Life expectancy more than 3 months
* Without EGFR-sensitive mutation (19Exon del/21Exon L858R), ALK, ROS1 gene rearrangement or fusion
* Has no prior systemic therapy; (chemotherapy and/or radiotherapy is allowed as part of neoadjuvant/adjuvant therapy. Patients who have had recurrence or metastasis for more than 6 months from the end of neoadjuvant/adjuvant treatment would be enrolled)
* ECOG score 0-1
* Patients must have at least one measurable lesion according to RECIST 1.1
* Has adequate organ function
* Agree to provide tumour tissue samples for biomarker exploration (including but not limited to PD-L1 IHC or NGS testing)
* Voluntarily sign a written informed consent form

Exclusion Criteria:

* Histological examination with Small Cell Lung Cancer or squamous Non-Small Cell Lung Cancer
* With active central nervous system (CNS) metastases confirmed by CT or MRI
* With other malignancy within 3 years before enrollment
* With severe infections within 4 weeks of the first dose of study treatment
* Women who are pregnant or lactating
* History of interstitial lung disease, drug-induced interstitial lung disease, or radiation pneumonia requiring hormone therapy
* History of myocarditis, cardiomyopathy, and malignant arrhythmia
* Tumor compresses important surrounding organs (such as the esophagus) with accompanying symptoms, compressing the superior vena cava or invading the mediastinal vessels, heart, etc.
* Risk of bleeding, major hemoptysis, or with history of coagulation dysfunction
* Active autoimmune diseases that require systematic treatment within 2 years before enrollment
* History of Human Immunodeficiency Virus (HIV)
* With active hepatitis B infection
* With uncontrollable pleural effusion, pericardial effusion, or ascites that require repeated drainage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
12-month progression-free-survival (PFS) rate | At 12 months
  Rate of patients with complete/partial response at 12-month from enrollment

SECONDARY OUTCOMES:
objective response rate (ORR) | about 24 months
  objective response rate using RECIST 1.1 criteria
duration of response (DOR) | about 24 months
  Time from the date of the first documented response (CR or PR) to the earliest date of disease progression (RECIST 1.1), or death due to any cause
disease control rate (DCR) | about 24 months
  disease control rate using RECIST 1.1 criteria
time to response (TTR) | about 24 months
  Time from the date of enrollment to the first documented response (CR or PR) (RECIST 1.1)
progression free survival (PFS) | about 24 months
  Time from enrollment to first observation of progression (RECIST1.1) or date of death (from any cause)
overall survival (OS) | about 24 months
  Time from enrollment until death due to any cause
incidence, type and severity of adverse events | From time of informed consent through treatment period and up to 30 days post last dose of study treatment (about 24 months)
  Descriptive statistics of safety will be presented using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qian Chu, Principal Investigator — Tongji Hospital
Locations (1):
- Qian Chu, Wuhan, Hubei, China